CLINICAL TRIAL: NCT03679793
Title: A Prospective Randomized Comparative Study of Open and Percutaneous Release of Acquired Trigger Thumb
Brief Title: Study of Open and Percutaneous Release of Acquired Trigger Thumb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr TSE Wing Lim, Associate Consultant and Clinical Associate Professor (Honorary), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trigger thumb_Protocol_v02
Record Dates: First submitted 2018-09-03; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Trigger Thumb
Keywords: Trigger Finger Disorder; Trigger Thumb; Minimally Invasive Surgical Procedures; Orthopedics
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Release Group (Active Comparator): Open surgical release of the A1 pulley is the gold standard of treating symptomatic trigger finger.
  Interventions: Procedure: Open Release Group
- Percutaneous Release Group (Experimental): Percutaneous release is a minimal invasive alternative surgical procedure
  Interventions: Procedure: Percutaneous Release Group

INTERVENTIONS:
Procedure: Open Release Group — Open surgical release of the A1 pulley is the gold standard of treating symptomatic trigger finger
  Arms: Open Release Group
Procedure: Percutaneous Release Group — Percutaneous release is a minimal invasive alternative surgical procedure
  Arms: Percutaneous Release Group

SUMMARY:
Trigger finger, also known as trigger digit or stenosing tenovaginitis, is caused by a size mismatch between the flexor tendon and the A1 pulley, which is generally characterized by pain, swelling, the limitation of finger range of motion and a symptomatic locking or clicking sensation. Conservative treatment options include the application of non-steroidal anti-inflammatory drugs (NSAID), physiotherapy, electrotherapy, splinting and corticosteroid injection but not always effective with regard to frequent recurrence. Open surgical release of the A1 pulley remains the gold standard of treating symptomatic trigger finger. While percutaneous release is a minimal invasive alternative and gaining popularity for the index, middle ring and little fingers, investigations for the surgical efficacy on thumb is few and far between. Investigators believe that a carefully conducted operation with proper positioning of the thumb, wide-awake approach and meticulous technique can achieve similar efficacy and safety in terms of possibly less intraoperative pain, imperceptible scar and early return to daily activities and routine work.

The hypothesis of this study is that by using a proper positioning of thumb, wide awake approach and meticulous technique in conducting percutaneous release of trigger thumb can achieve similar efficacy and safety compared to that of open release surgical method. Moreover, percutaneous release of trigger thumb can generate less intraoperative pain, imperceptible scar and promote early return to routine work.

Hence, the objective of this study is to investigate and compare the safety, effectiveness and outcome of percutaneous release versus traditional open release for trigger thumbs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of trigger thumb with Green's staging graded 2-4
* Patients were unresponsive to conservative treatments for more than 3 months (Nonsteroidal anti-inflammatory drugs, physiotherapy, splinting, or injection of steroid)

Exclusion Criteria:

* With history in rheumatoid arthritis
* Unable to give verbal or written consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Total volume of local anaesthetics injected | Intra-operative
  The total volume of local anaesthetics injected during operation
Duration of surgery (in minutes) | Intra-operative
  The time (in minutes) needed for operation
Surgical site pain | Intra-operative
  Visual analogue scale (VAS) was used to evaluate the pain at surgical site (0=no pain and 10=greatest pain)
Active and passive range of motion (ROM) of interphalangeal joint (IPJ) and metacarpal-phalangeal joint (MPJ) | Pre-operative
  Pre-operative active and passive ROM of IPJ and MPJ was measured to determine the joint stiffness
Active and passive range of motion (ROM) of interphalangeal joint (IPJ) and metacarpal-phalangeal joint (MPJ) | Post-op Day 7
  Active and passive ROM of IPJ and MPJ was measured post-operatively to determine the joint stiffness
Active and passive range of motion (ROM) of interphalangeal joint (IPJ) and metacarpal-phalangeal joint (MPJ) | Post-op Day 28
  Active and passive ROM of IPJ and MPJ was measured post-operatively to determine the joint stiffness
Active and passive range of motion (ROM) of interphalangeal joint (IPJ) and metacarpal-phalangeal joint (MPJ) | Post-op Day 90
  Active and passive ROM of IPJ and MPJ was measured post-operatively to determine the joint stiffness
Pre-operative Kapandji score | Pre-operative
  Kapandji score is a tool useful for assessing the opposition of the thumb, based on where on their hand the patient is able to touch with the tip of their thumb.
Post-operative Kapandi score | Post-op Day 7
  Kapandji score is a tool useful for assessing the opposition of the thumb, based on where on their hand the patient is able to touch with the tip of their thumb.
Post-operative Kapandi score | Post-op Day 28
  Kapandji score is a tool useful for assessing the opposition of the thumb, based on where on their hand the patient is able to touch with the tip of their thumb.
Post-operative Kapandi score | Post-op Day 90
  Kapandji score is a tool useful for assessing the opposition of the thumb, based on where on their hand the patient is able to touch with the tip of their thumb.
Pre-operative Disabilities of the Arm, Shoulder and Hand (DASH) scores, including total, function, symptoms and work | Pre-operative
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
Post-operative Disabilities of the Arm, Shoulder and Hand (DASH) scores, including total, function, symptoms and work | Post-op Day 7
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
Post-operative Disabilities of the Arm, Shoulder and Hand (DASH) scores, including total, function, symptoms and work | Post-op Day 28
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
Post-operative Disabilities of the Arm, Shoulder and Hand (DASH) scores, including total, function, symptoms and work | Post-op Day 90
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
Pre-operative pain at rest | Pre-opeartively
  Visual analogue scale (VAS) was used to evaluate the pain at rest (0=no pain, 10=greatest pain)
Post-operative pain at rest | Post-op Day 7
  Visual analogue scale (VAS) was used to evaluate the pain at rest (0=no pain, 10=greatest pain)
Post-operative pain at rest | Post-op Day 28
  Visual analogue scale (VAS) was used to evaluate the pain at rest (0=no pain, 10=greatest pain)
Post-operative pain at rest | Post-op Day 90
  Visual analogue scale (VAS) was used to evaluate the pain at rest (0=no pain, 10=greatest pain)
Pre-operative pain on exertion | Pre-operative
  Visual analogue scale (VAS) was used to evaluate the pain on exertion (0=no pain, 10=greatest pain)
Post-operative pain on exertion | Post-op Day 7
  Visual analogue scale (VAS) was used to evaluate the pain on exertion (0=no pain, 10=greatest pain)
Post-operative pain on exertion | Post-op Day 28
  Visual analogue scale (VAS) was used to evaluate the pain on exertion (0=no pain, 10=greatest pain)
Post-operative pain on exertion | Post-op Day 90
  Visual analogue scale (VAS) was used to evaluate the pain on exertion (0=no pain, 10=greatest pain)
Satisfaction level after surgery | Post-op Day 7
  Subjects' satisfaction was evaluated (1=totally not satisfied; 10=totally satisfied) after surgery
Satisfaction level after surgery | Post-op Day 28
  Subjects' satisfaction was evaluated (1=totally not satisfied; 10=totally satisfied) after surgery
Satisfaction level after surgery | Post-op Day 91
  Subjects' satisfaction was evaluated (1=totally not satisfied; 10=totally satisfied) after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics and Traumatology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
All collected data were from patients from study site and strictly confidential